CLINICAL TRIAL: NCT05372289
Title: Immunonnutrition in Spine Surgery to Improve Patient's Outcome: a Randomized Controlled Trial
Brief Title: Preoperative Immunonutrition in Patients Undergoing Spine Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ORTHOPACT (PI: M Briguglio); L4144 (Other Grant/Funding Number: Italian Ministry of Health)
Record Dates: First submitted 2022-05-09; First posted 2022-05-12 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Arthrosis; Spine
MeSH Terms: conditions — Osteoarthritis | interventions — Immunonutrition Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: In this study, the primary endpoint assessors, who are assessing parameters constituting the primary endpoints, will be masked to the treatment regimen. Any personnel involved with the statistical analysis and interpretation of the data and results will be masked to the treatment regimen until database lock.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplemented patients (Experimental)
  Interventions: Dietary Supplement: Immuno-nutrition
- Standard of care (No Intervention)

INTERVENTIONS:
Dietary Supplement: Immuno-nutrition — The experimental group of 68 older adults will be subjected to a preoperative immuno-nutrition for 30 days prior to surgery and up to 3 days after surgery. The oral feed provides energy, omega-3 fatty acids, arginine, nucleotides, and soluble fibre.
  Arms: Supplemented patients

SUMMARY:
A malnutritional status is known to be associated with altered immune function, reduced function, and worsen outcomes after orthopedic surgery. Medical and surgical complications are not uncommon in Orthopedics and infection rates are potentially life-threatening complications, with the highest morbidity, mortality, and healthcare costs. Most patients undergoing orthopedic surgery are elderly, malnourished, osteosarcopenic, sedentary, anemic, and suffer from low levels of vitamin D. A mono-nutrient supplement may be not sufficient for supporting the arthrodesis techniques, which are invasive open surgeries procedures with significant blood losses and the need of transfusions. In this therapeutic area, immuno-nutrition has been used in spine surgery, with the reduction of complications, revisions, and readmissions. In addition, prosthetic surgery outcomes have been observed to ameliorate by using this nutritional support. Therefore, preoperative oral immuno-nutrition therapy may be applied in older adults undergoing spine surgery to improve patients' outcomes and reduce complications.

This is a randomized, controlled, open-label, 2-arm non-parallel-group, single-center interventional study to assess the efficacy of an immuno-nutrition therapy vs. hospital standard of care in spine surgery to improve patients' outcomes. This is a single primary endpoint study. A total of 136 patients from IRCCS Orthopedic Institute Galeazzi in Italy will be recruited and assigned in a 1:1 ratio to the treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* male and female sex, of all ethnicities, aged over 60
* arthrodesis involving ≥ 6 vertebrae
* American Society of Anesthesiology (ASA) risk: 1, 2, or 3
* Absence of neurological or psychiatric disorders
* Signing of informed consent and consent to collaborate in all study procedures
* Patients who meet the clinical requirements to undergo their first spinal surgery

Exclusion Criteria:

* American Society of Anesthesiology (ASA) risk: 4
* No cervical arthrodesis
* Diagnosis of neurological or psychiatric disorders
* Revisions
* Therapy with other supplements at the time of the first visit 0
* Known allergy or adverse food reactions
* Chronic inflammatory or autoimmune diseases (e.g. rheumatoid arthritis)
* Gastrointestinal disorders
* Conditions that do not allow to undergo surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2022-03-16 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Amelioration of functions evaluated through the Oswestry Disability Index (ODI) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Briguglio, Principal Investigator — IRCCS Istituto Ortopedico Galeazzi
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided